CLINICAL TRIAL: NCT05937035
Title: Histological and Volumetric Evaluation of Customized Allograft Bone Blocks in Severe Atrophy of the Mandible: a Prospective Cohort Clinical Trial
Brief Title: Histological and Volumetric Evaluation of Customized Allograft Bone Blocks
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat Internacional de Catalunya (Other)
Responsible Party: Principal Investigator, Jordi Gargallo-Albiol, MD, PhD Prof., Universitat Internacional de Catalunya
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIR-ECL-2022-02
Record Dates: First submitted 2023-05-09; First posted 2023-07-10 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Alveolar Bone Resorption; Graft Overgrowth; Resorption of Bone Graft; Graft Complication; Block
MeSH Terms: conditions — Bites and Stings

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Customized allogenic bone block (Other): 1 group to study
  Interventions: Procedure: Customized allogenic bone block surgery

INTERVENTIONS:
Procedure: Customized allogenic bone block surgery — After studying the CBCT to regenerate the posterior sites of the mandible, the investigators will design CAD/CAM freeze- dried bone allograft to fit exactly on the defect morphology that the patients present. A full thickness flap will be released to have a correct access of the defects. Releasing incisions will be performed to achieve the correct closure of the flap. The sterile blocks have to fit perfectly on the defect and fixed by screws. Covered with resorbable membranes fixed with pines and suture. 4 months later, photographs, periapical xrays digital impressions and 2nd CBCTwill be performed. During the implant surgery, a bone trephine will be removed and sent into a Laboratory to make a histological study of the bone block for histomorphometry. After 3 months, second-stage surgery and healing caps will be placed if needed. Impressions will be taken 2 weeks after to perform the final crowns.

SUMMARY:
Customized bone blocks need CBCT and digital software to design the block needed to rehabilitate. Some advantages are reduced surgical time and better adaptation of the graft, leading to less complications.

Objectives: The primary aim of this study is to determine the bone regeneration capacity through a histological study and the bone volumetric changes of allograft bone blocks in the posterior site of the mandible. The secondary outcome will be to assess the survival and success rate of dental implants placed in the allograft regenerated area.

Materials and Methods: After studying the CBCT to regenerate the posterior sites of the mandible, the investigators will design CAD/CAM freeze- dried bone allograft to fit exactly on the defect morphology that the patients present. A full thickness flap will be released to have a correct access of the defects. The sterile blocks have to fit perfectly on the defect and fixed by screws. Covered with resorbable membranes fixed with pines and suture. 4 months later, 2nd CBCTwill be performed. During the implant surgery, a bone trephine will be removed and sent into a Laboratory to make a histological study of the bone block for histomorphometry. After 3 months, second-stage surgery and healing caps will be placed if needed. Impressions will be taken 2 weeks after to perform the final crowns.

DETAILED DESCRIPTION:
Allogenic bone blocks are a great bone regeneration technique option comparing to autologous regeneration treatments. There are several techniques of vertical guided bone regeneration but also have a large number of complications and failures. Some of the advantages of Customized Allograft Bone Blocks are: less invasive, causes less morbidity and resorption of the recipient site. Non resorbable membranes with particulate grafting material and autologous bone blocks are technically demanding and difficult to achieve stability to create new bone. Customized bone blocks need CBCT and digital software to design the block needed to rehabilitate. It is important to place the implants in an ideal prosthetic position to achieve excellent long-term results. Implant supported prosthesis can be contraindicated because of the lack of bone. Looking in to the classification of CAWOOD and HOWEL type 5 bone need bone augmentation techniques. In some cases, increasing the difficulty with the superficialization of the alveolar nerve. Some advantages are reduced surgical time and better adaptation of the graft, leading to less complications. The use of autogenous bone increases the risk of damaging anatomical structures increasing the morbidity, however thanks to allograft the investigators can avoid these problems. There are many different types of allografts, fresh-frozen bone (FFBA), freeze-dried bone (FDBA), demineralised freeze-dried bone allograft (DFDBA) and mineralised processed bone (MPBA). The allograft used for this study is a cellular cancellous bone material mechanically and chemically processed and sterilised by irradiation. This allogenic biomaterial has an osteoconductive property which facilitates the cell migration and proliferation for neoformation.

Study design A prospective controlled clinical trial will be conducted.

Residents of the International Master in Oral Surgery will perform the surgical and prosthodontic final rehabilitation procedures. All the included patients will sign an appropriate inform prior to any study-related actions. Firstly, an intraoral digital impression with intraoral scanner will be taken and a diagnostic wax-up will be performed. Subsequently, a cone-beam computed tomography scan would be taken in the specific area to be treated. After studying the CBCT to regenerate the posterior sites of the mandible, the investigators will design CAD/CAM freeze- dried bone allograft to fit exactly on the defect morphology that the patients present. A full thickness flap will be released to have a correct access of the defects. Releasing incisions will be performed to achieve the correct closure of the flap. The sterile blocks have to fit perfectly on the defect and fixed by screws. Covered with resorbable membranes fixed with pines and suture. 4 months later, photographs, periapical xrays digital impressions and 2nd CBCT will be performed. During the implant surgery, a bone trephine will be removed and sent into a Laboratory to make a histological study of the bone block for histomorphometry. After 3 months, second-stage surgery and healing caps will be placed if needed. Impressions will be taken 2 weeks after to perform the final crowns.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent
2. Overall, healthy subjects (ASA1 and 2)
3. Females and males of at least eighteen-years
4. Requiring a posterior mandible rehabilitation with a minimum of 2 dental implants
5. Able to follow instructions and attend a regular compliance

Exclusion Criteria:

1. Acute local infection
2. Untreated periodontal disease assessed by Socransky et al. parameters (≥ 2mm clinical attachment loss in two consecutive visits within 1 year)
3. Drug and/or alcoholic dependencies
4. Medical conditions contraindicating implant surgery
5. History of head and/or neck radiation
6. Bisphosphonate therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-05-25 (Estimated); Primary Completion 2024-09-25 (Estimated); Study Completion 2025-07-25 (Estimated)

PRIMARY OUTCOMES:
Histological study | 2 years
  histological study (histological analysis). Histomorphometry analysis will be performed at 5 months during the implant placement surgery.
Bone volumetric changes | 2 years
  The bone volumetric changes of allograft bone blocks in the posterior site of the mandible. To assess the bone changes before and after implant treatment, CBCT scans are taken before bone regeneration, before implant placement at 4 months and 12 months after bone regeneration (Heigh and width) (mm)

SECONDARY OUTCOMES:
Survival rate of dental implants | 2 years
  Survival rate of dental implants placed in the allograft regenerated area (implants % survival)
Success rate | 2 years
  Success rate of dental implants placed in the allograft regenerated area (implants without complications after 2 yerars)
Complications | 2 years
  Evaluate the number of complications associated to this technique (%)

CONTACTS AND LOCATIONS:
Overall Officials: JORDI GARGALLO-ALBIOL, Principal Investigator — Universitat Internacional de Catalunya
Locations (1):
- Universitat Internacional de Catalunya, Sant Cugat del Vallès, Barcelona, Spain